CLINICAL TRIAL: NCT03878459
Title: Can Addition of Pioglitazone to SGLT2 Inhibitor in Type 1 Diabetic Patients Amplify the Decrease in HbA1c and Prevent the Increase in Plasma Ketone Concentration?
Brief Title: Dapagliflozin Plus Pioglitazone in T1DM
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC20180515H
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: T1DM,ketoacidosis, dapagliflozin, pioglitazone
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Pioglitazone

STUDY DESIGN:
Intervention Model Description: placebo controlled intervention
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): pioglitazone treatment
  Interventions: Drug: Pioglitazone 45 mg
- control (Placebo Comparator): subjects will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone 45 mg — patients will be started on 15 mg and the dose escalated to the maximal tolerated dose
  Arms: Intervention
Drug: Placebo — PATIENTS WILL RECEIVE PLACEBO
  Arms: control

SUMMARY:
Purpose: To examine the effect of addition of combination therapy with dapagliflozin plus pioglitazone to insulin on glucose control and plasma ketone concentration in patients with type 1 diabetes (T1DM) Research Design: 120 patients with type 1 diabetes who otherwise are healthy constitute the study population. After screening, eligible subjects will start 4 week run in. At week 4, subjects will receive dapagliflozin for 12 weeks. At week 16, subjects will be randomized to receive in a double blind fashion pioglitazone or placebo for 16 weeks.

Methods: the following techniques will be employed in the present study: (1) mixed meal tolerance test; (2) indirect calorimetry; (3) continuous glucose monitoring.

Clinical Relevance: the results of the present study will demonstrate that the addition of pioglitazone to SGLT2 inhibitor in T1DM patients produces greater reduction in the HbA1c without increasing risk of ketoacidosis and hypoglycemia.

DETAILED DESCRIPTION:
Insulin deficiency, due to autoimmune destruction of beta cells, is the primary factor responsible for the development of T1DM, and insulin replacement therapy is the mainstay for the management of hyperglycemia. However, insulin therapy often is associated with adverse events, including weight gain which promotes insulin resistance leading to an increase in insulin demand. This results in a self-perpetuating vicious cycle whereby the increase in insulin dose causes weight gain that worsens insulin sensitivity, and further enhances insulin requirement. Hyperinsulinemia per se also induces insulin resistance.

To break this cycle, adjunctive therapies have been added to insulin in T1DM patients to lower the plasma glucose concentration. However, the addition of metformin, pioglitazone, and GLP-1 agonists to insulin in T1DM patients have not provided convincing evidence for a clinically meaningful reduction in the HbA1c or significant reduction in daily insulin dose.

SGLT2 inhibitors (SGLT2i) are a novel class of antidiabetic agents which reduce the plasma glucose concentration by inhibiting renal glucose reuptake and producing glucosuria. Because of this unique mechanism of action, which is independent of insulin secretion and insulin action, SGLT2i have proven to be very effective in lowering the plasma glucose concentration in T1DM. Initial proof of concept studies have demonstrated that, compared to placebo, all members of this class (dapagliflozin, empagliflozin, canagliflozin and sotagliflozin) effectively lower the plasma glucose concentration, HbA1c and daily insulin dose in T1DM without increased risk of hypoglycemia. Further, SGLT2i improved cardiovascular risk factors in T1DM by promoting weight loss and decreasing blood pressure.

Despite the promising potential for SGLT2i as adjunctive therapy to insulin in T1DM, recent large clinical trials have demonstrated two important limitations to this therapeutic strategy: First, although the decrease in HbA1c caused by SGLT2i in T1DM patients was statistically significant, the absolute decrease was relatively modest (0.30-0.45%). The investigators, previously have shown that SGLT2i stimulate an increase in the basal rate of hepatic glucose production (HGP) in T2DM patients. This SGLT2i-induced increase in HGP offsets by approximately one half the amount of glucose lost in the urine. Therefore, the investigators have hypothesize that, similar to what they have observed in T2DM patients, the addition of SGLT2i to insulin in T1DM patients stimulates HGP thereby attenuating the decrease in HbA1c. Further, the decrease in daily insulin dose after initiating therapy with SGLT2i in T1DM patients would be expected to enhance the increase in HGP and diminish the decrease in HbA1c. Thus, preventing the increase in HGP caused by SGLT2i in T1DM can be expected to markedly amplify the clinical efficacy of SGLT2i and enhance the reduction in HbA1c.

A second limitation of the use of SGLT2i an adjunct therapy to insulin in T1DM patients is the increase in diabetic ketoacidosis (DKA) risk. In three large clinical trials , the addition of SGLT2i to insulin in T1DM patients was associated with a 3-6% increase in DKA risk (see Table 1 below). Because of the significant morbidity and mortality associated with DKA, the increased DKA risk in T1DM has raised concerns about the use of SGLT2i as an adjunct therapy to insulin in T1DM patients despite their multiple metabolic benefits.

The Investigators previously have demonstrated that SGLT2i cause a significant increase in plasma FFA concentration, fat oxidation and subsequent increase in plasma ketone concentration in T2DM patients (27). Therefore, they hypothesize that in T1DM, SGLT2i cause a similar increase in plasma FFA concentration, fat oxidation and plasma ketone concentration which in certain clinical conditions (e.g. acute illness) can increase the production of ketones and result in the development of DKA. Further, prevention of the increase in plasma FFA concentration will inhibit the increase in plasma ketone concentration and reduce DKA risk associated with SGLT2i use in T1DM patients.

Pioglitazone inhibits lipolysis and markedly decreases the plasma FFA concentration. Further, pioglitazone is a potent inhibitor of HGP. These actions of pioglitazone are due to direct actions of the drug on adipocytes and liver, respectively, are mediated by PPAR gama, and are independent of the plasma insulin and glucagon concentrations. In fact, pioglitazone inhibits lipolysis and HGP in type 2 diabetic patients despite a decrease in plasma insulin concentration. Therefore, the investigators hypothesize that the addition of pioglitazone to SGLT2i in T1DM patients will prevent the rise in HGP caused by SGLT2i and, thereby, augment the decrease in HbA1c. Further, combination therapy with pioglitazone plus SGLT2i will prevent the increase in plasma FFA concentration and subsequent increase in plasma ketone concentration, thus reducing the risk of DKA.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* T1DM
* Good general health
* Fasting C-peptide concentration <0.7 ng/ml
* Poor glycemic control (HbA1c=7.0-11.0%)
* Treatment with multiple daily insulin injections or insulin pump
* Total daily insulin dose ≥0.6 U/kg per day
* Stable insulin dose (±4 units) in the preceding three months.
* eGFR≥60 ml/min
* Weight stable over the preceding 3 months (± 3 pounds)
* Do not participate in an excessively heavy exercise program

Exclusion Criteria:

* T2DM
* Daily insulin dose <0.6 U/kg per day
* Fasting C-peptide >0.7 ng/ml
* HbA1c <7.0% or >11.0%
* eGFR<60 ml/min
* Hematuria in urine analysis
* Pregnancy, lactating, positive pregnancy test or planning to become pregnant in the following year.
* Women of child-bearing potential will be requested to use at least two barrier methods before being enrolled in the study.
* Major organ system disease which includes: (i) malignancy or history of malignancy including bladder cancer; (ii) Congestive heart failure or history of coronary heart disease or any other cardiac disease; (iii) chronic liver disease or LFT >3 times the upper normal level; (iv) History of alcohol or drug abuse; (v) History of chronic lung disease (e.g., COPD, asthma); (vi) history of rheumatic disease; (vii) History of chronic pancreatitis or pancreatic surgery; (viii) History of CVA or TIA (ix) Planned surgery during the study; (x) history of HIV infection or other immune compromised disease; and history of organ transplantation; (xi) patients who take medications, other than insulin, known to affect glucose metabolism, e.g., prednisone.
* Evidence of proliferative diabetic retinopathy
* Patients enrolled in a heavy exercise program
* Patients on ketogenic diet
* History of hospitalization for DKA, hypoglycemia or uncontrolled hyperglycemia in the preceding 6 month.
* Presence of symptoms of poor glycemic control, e.g. polydipsia or polyurea
* History of hypersensitivity to dapagliflozin or pioglitazone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-08-08 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Decrease in HbA1c | 28 weeks

SECONDARY OUTCOMES:
plasma ketones | 28 weeks
  increase in plasma ketone concentration
insulin dose | 28 weeks
  decrease in daily insulin dose

CONTACTS AND LOCATIONS:
Locations (3):
- University Health System Texas Diabetic Institute, San Antonio, Texas, United States
- Endocrinology and Diabetes Center, Rambam Medical Center, Haifa, Israel
- Dasman Diabetes Institute, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: No